CLINICAL TRIAL: NCT00002009
Title: A Phase I/II Study of Recombinant Human GM-CSF in Patients With AIDS Virus Infection and Leukopenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 067E; 101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1988-06

CONDITIONS: HIV Infections; Cytopenias
Keywords: Leukopenia; Drug Evaluation; Granulocyte-Macrophage Colony-Stimulating Factor
MeSH Terms: conditions — HIV Infections; Cytopenia; Leukopenia | interventions — sargramostim

INTERVENTIONS:
Drug: Sargramostim

SUMMARY:
To determine the maximum tolerated dose (MTD) and toxicity of sargramostim (recombinant granulocyte-macrophage colony-stimulating factor; GM-CSF) given by continuous intravenous infusion (CIV) in patients with leukopenia in association with AIDS virus infection. In addition, single dose and steady state pharmacokinetics will also be determined.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Met the CDC criteria for the diagnosis of AIDS.
* Total peripheral blood leukocyte count = or < 3000 cells/mm3 measured on at least two occasions separated by a minimum of one week.
* Must have or have recovered from one or more opportunistic infection.
* Serum antibody to HTLV-III/LAV with or without viremia.
* Anticipated survival of at least 6 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* AIDS related complex (ARC).
* History of malignancy other than Kaposi's sarcoma (KS).
* Excessive diarrhea (more than 5 liquid or non-liquid stools per day).
* Currently hospitalized or hospitalized within the last 4 weeks for the treatment of opportunistic infections.
* Presence of renal dysfunction.
* Other evidence of primary hematologic or infectious disorders unrelated to AIDS virus infection.

Patients with the following are excluded:

* AIDS related complex (ARC).
* History of malignancy other than Kaposi's sarcoma (KS).
* Excessive diarrhea (more than 5 liquid or non-liquid stools per day).
* Currently hospitalized or hospitalized within the last 4 weeks for the treatment of an opportunistic infection.
* Dementia or altered mental status that would prohibit the giving and understanding of informed consent.

Prior Medication:

Excluded:

* Any marrow suppressive medications such as trimethoprim-sulfamethoxazole combination (TMP-PurposeX) or Fansidar.
* Excluded within 6 weeks of study entry:
* Any investigational drug.

Prior Treatment:

Excluded within 6 weeks of study entry:

* Systemic cytotoxic chemotherapy or irradiation.

Risk Behavior:

Excluded within 3 months of study entry:

* Regular, excessive use of alcohol, hallucinogens or agents which are addicting.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA CARE Ctr, Los Angeles, California
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts

REFERENCES:
- [Background] Barbarini G, Garavelli G, Grisorio B, Barbaro G, Giangregorio F. GM-CSF in HIV related leukopenia: efficacy and tolerability of three months therapy on 50 patients. Int Conf AIDS. 1996 Jul 7-12;11(1):313 (abstract no TuB2279)